CLINICAL TRIAL: NCT03750838
Title: Refining and Piloting a Text Messaging Intervention to Delay Alcohol Initiation and Reduce Alcohol Use Escalation Among Abstainer and Lighter Drinker College Students
Brief Title: Alcohol Intervention for First Year College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Dana Litt, PhD., Associate Professor of Health Behavior and Health Systems, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA026004 (NIH); 1R34AA026004-01A1 (NIH)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Underage Alcohol Use
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Messaging Intervention Group (Experimental): Participants in the Text Messaging Intervention condition will be provided a predetermined number of messages per week (based partially on responses from Phase 2 focus group) for 6 weeks delivered on Thursdays, Fridays, and Saturdays, which are the most common days of the week that heavy drinking occurs as well as other days and times that focus group participants indicated would be the most helpful.
  Interventions: Behavioral: Text Messaging Intervention
- Assessment Only Control (No Intervention): Participants in the assessment only control will not receive any text messages, but will complete all survey assessments on the same schedule as the Text Message Intervention Group.

INTERVENTIONS:
Behavioral: Text Messaging Intervention — The content for the text messaging Intervention will be designed to be non-confrontational in tone, seek to increase motivation to drink lightly or not at all, and based both on general information about light and non-drinking as well as information provided during the baseline assessment.
  Arms: Text Messaging Intervention Group

SUMMARY:
While a large focus of research on U.S. college drinking has focused on the prevalence of and problems related to heavy-episodic drinking, less has focused on college students who are either abstainers or lighter drinkers (i.e., for men, drinking 4 or fewer drinks in two hours and 14 or fewer drinks per week; and for women drinking 3 or fewer in two hours and 7 or fewer drinks per week). Over 40% percent of college students ages 18-22 do not report drinking in the past month with only half of those engaging in regular heavy-episodic drinking. Research suggests that a significant proportion of students who were abstinent or light drinkers prior to and upon entering college initiate drinking and progress to becoming heavy-episodic drinkers. This provides evidence that the first few months of college is a high-risk time for initiating both drinking and heavy-episodic drinking and that delaying the onset of heavy-episodic drinking among light drinkers and abstainers should lead to reduced harms throughout the college years and young adulthood. Mobile phone-based interventions are an innovative method for reaching young people and have been established as an empirical approach towards addressing health issues, including alcohol use. The ultimate goal of this proposal is to develop, refine and pilot a text message (TM) intervention for abstainer and lighter drinking first year college students with the ultimate goal of delaying alcohol initiation and/or reducing alcohol use escalation. An iterative process of focus groups, intervention content development, and user feedback focused on the unique experiences of abstainers and lighter drinkers will inform the TM Intervention to be delivered in a pilot study with 6 weeks of TMs. The pilot study will include a 6 week post-intervention assessment, and 3, 6, and 9 month follow-ups among 100 incoming first year abstainer and lighter drinker college students. Given that reducing young adults' and college students' engagement in excessive alcohol use has been listed as a major objective of Healthy People 2020 and a key priority of NIAAA, an intervention that focuses on delaying alcohol initiation and escalation into higher-risk alcohol use among abstainer and lighter drinkers could make important strides to achieving this goal.

DETAILED DESCRIPTION:
The first year at college, and specifically the first 6 weeks of college, has been identified as a critical period particularly influential to college students' alcohol use trajectories. The prevalence of heavy drinking increases rapidly upon college entry relative to pre-college use and patterns of high-risk alcohol use established during the transition to college can result in a range of adverse consequences that persist throughout the academic year. While a large focus of research on U.S. college drinking has been on the prevalence of and problems related to heavy-episodic drinking (4+/5+ drinks in two hours for women/men), less research has focused on college students who are either abstainers (i.e., do not drink any alcohol) or lighter drinkers (i.e., men: 4 or fewer drinks in two hours and 14 or fewer drinks per week; women: 3 or fewer in two hours and 7 or fewer drinks per week). Research indicates that between 21% and 26% of first-year colleges students who were abstinent or light drinkers before college escalated to heavy episodic drinking during their freshman year. Further, over 40% percent of college students ages 18-22 do not report drinking in the past month, with only half of those engaging in regular heavy-episodic drinking. Research indicates that risk cognitions (i.e., prototypes, norms) are associated with initiation and escalation of alcohol use and also tend to peak around the time that individuals transition out of high school and into a riskier college environment. Delaying the onset of heavy-episodic drinking among abstainers and lighter drinkers during the first-year of college, a particularly high-risk period, should lead to reduced related harms throughout both the college years and young adulthood.

Tailoring intervention approaches to students at various levels of risk, including abstainers or lighter drinkers, may greatly increase efficacy and reduce costs associated with universal interventions (King et al., 2008). No single intervention is likely to sufficiently reduce college drinking or consequences; therefore a "mix of strategies is best". An underexplored strategy is delivering intervention content that reinforces existing reasons for not drinking among abstainers and lighter drinkers, with the goal of delaying the initiation of heavy drinking and/or the escalation to heavy drinking during the first year of college. Given that longitudinal findings indicate that stronger endorsement of reasons for drinking lightly or not drinking, such as academic responsibilities, normative influence, and concern for social images are associated with delayed alcohol initiation, lower levels of alcohol use and higher rates of abstention among young adults, including college students, interventions for abstainers and lighter drinkers that focus on reinforcing proximal reasons not to drink or to drink lightly have promise to dissuade students from initiation of drinking or to delay more hazardous drinking patterns later on.

Additionally, mobile phone-based interventions are an innovative method for reaching young people and have been established as an evidence-based, recommended approach towards addressing health issues including alcohol use. Mobile phone text-messaging (TM) offers an innovative technological approach to brief intervention for college students in a mode in which they are familiar and they already use frequently. Presenting preventative intervention content via TM, especially for abstainer and lighter drinking college students, may be one way to delay alcohol use initiation and prevent the escalation of alcohol use during the first year of college. Therefore, the present project has the following primary aims:

Aim 1: Recruit first year college students who are abstainers and lighter drinkers to examine students' reactions to TM intervention content through an iterative process of focus groups, intervention content development, and user feedback, which will inform a new intervention to be delivered in a pilot study (Aim 3).

Aim 2: Through focus groups, elicit responses to timing of the TM intervention, specifically what days and times per week and how many times per day (set within research-established ranges) abstainer and lighter drinkers think receiving TMs will the most useful and impactful to inform TM delivery for the pilot study (Aim 3).

Aim 3: Conduct a pilot study with 6 weeks of TM intervention content, a 6 week post-intervention assessment and 3, 6, and 9 month follow-ups among 100 abstainer or lighter drinking first-year college students to determine feasibility, acceptability, and preliminary effect sizes (to estimate power and sample sizes for a future R01). Newly enrolled first-year college students will be randomized to the TM intervention or assessment only control. The investigators hypothesize the TM Intervention will be feasible and acceptable to abstainer and lighter drinking students, including being accessible, usable, convenient, relevant and helpful. The investigators further hypothesize that receiving the TM intervention will be associated with less initiation and escalation of drinking, fewer negative consequences, more favorable prototypes of abstainers and lighter drinkers, greater perceived abstaining and light drinking norms, greater engagement and enjoyment of alternative activities, and greater endorsement of personal goals that do not involve alcohol at the 6 week post-intervention assessment and 3, 6, and 9 month follow-ups relative to assessment only control.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria includes:

* age 18-19 (see Identity and Age Verification below; If a participant screens in at 18 and turns 20 prior to the focus group, the participant will be allowed to be in the research study.)
* birth date that is consistent with their given age
* first-year college student at the University of North Texas
* valid email address
* have a text messaging plan on their mobile phone
* drinking 14/7 or fewer drinks per week for men/women
* no episodes in the past month of consuming 5/4 drinks in two hours for men/women
* express any willingness to take a sip of alcohol
* if female, must not be pregnant or trying to get pregnant
* willing to participate in focus groups at the University of North Texas

Exclusion Criteria:

* Not meeting inclusion criteria
* unwillingness to participate
* failure to provide consent (e.g., declining participation in the study)
* providing inconsistent responses (e.g., age) identified by the survey
* having already participated in the study as identified by overlap or consistency in computer IP addresses, contact information, and demographics

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 99 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Litt, PhD., Principal Investigator — University of North Texas Health Science Center
Locations (1):
- Dana, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
A select number of researchers will have access to unidentified participant data at the close of the study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Campus including in-person recruitment (e.g., tabling, distributing flyers at dorms), online recruitment, and sending student directory email invitations. Flyers advertising recruitment for the study were distributed at the on-campus orientation events and in student dorms with general, brief information about the study, links (URL and QR codes) to the screening survey, and the study's email address, and phone number. We recruited participants from June- August 2021.
Pre-assignment Details: Participants who were eligible, but did not complete the baseline survey were not fully enrolled and randomized to condition.
Groups:
- Text Messaging Intervention Group: Participants in the Text Message Intervention condition will be provided a predetermined number of messages per week (based partially on responses from Phase 2 focus group) for 6 weeks delivered on Thursdays, Fridays, and Saturdays, which are the most common days of the week that heavy drinking occurs as well as other days and times that focus group participants indicated would be the most helpful.
  Text Messaging Intervention: The content for the Text Message Intervention will be designed to be non-confrontational in tone, seek to increase motivation to drink lightly or not at all, and based both on general information about light and non-drinking as well as information provided during the baseline assessment.
- Assessment Only Control: Participants in the assessment only control condition completed all assessments on the same schedule as the Text Message Intervention group, but dot receive any text messages.
Period: Overall Study
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Started | 49 | 50
6 Week Follow-up | 40 | 43
3 Month Follow-up | 32 | 40
6 Month Follow-up | 37 | 44
Completed (9 month follow-up) | 39 | 44
Not Completed | 10 | 6
Not completed — Lost to Follow-up | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Text Messaging Intervention Group: Participants in the TM Intervention condition will be provided a predetermined number of messages per week (based partially on responses from Phase 2 focus group) for 6 weeks delivered on Thursdays, Fridays, and Saturdays, which are the most common days of the week that heavy drinking occurs as well as other days and times that focus group participants indicated would be the most helpful.
  Text Messaging Intervention: The content for the TM Intervention will be designed to be non-confrontational in tone, seek to increase motivation to drink lightly or not at all, and based both on general information about light and non-drinking as well as information provided during the baseline assessment.
- Active Control: Participants in the attention only control condition will receive a series of TM based on nutritional data on the same schedule as those in the TM intervention and will complete a 6 week post-intervention assessment as well as all follow-ups.
  Active Control: Participants will receive a series of TM based on nutritional data on the same schedule as those in the TM intervention and will complete a 6 week post-intervention assessment as well as all follow-ups.
- Total: Total of all reporting groups
Arm/Group | Text Messaging Intervention Group | Active Control | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 50 | 99
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.06 (0.24) | 18.12 (0.33) | 18.09 (0.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 35
  Not Hispanic or Latino | 33 | 30 | 63
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 23 | 35 | 58
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
Current Non-Drinkers [Count of Participants; unit: Participants] — Number of participants who do not currently drink alcohol at baseline.
  Participants | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Acceptability-Number of Participants Who Found the Study Overall Favorable
Description: Item assessing whether participants found the study overall favorable as measured at 6-week follow-up.
Time Frame: 6 weeks
Population: Acceptability data only collected from intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 40 | 0
Participants | 38 | 0

2. Primary Outcome: Acceptability-proportion of Participants Who Would Recommend the Study
Description: Item assessed by asking whether participants would recommend the study to other first-year college students
Time Frame: 6 weeks
Population: Only those participants assigned to intervention were shown these items.
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 40 | 0
Participants | 36 | 0

3. Primary Outcome: Acceptability and Feasibility-ratings of Text Message Content Areas
Description: Text Message Rating Scale- assessed ratings of text message intervention content areas with a minimum value of 0 and a maximum value of 4 with higher numbers being a better outcome (i.e., more acceptable)
Time Frame: 6 weeks
Population: Acceptability was only measured for those in text message intervention group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 24 | 0
units on a scale
  Substance free activities text messages | 3.27 (0.16) |
  Image text messages | 3.00 (0.47) |
  Norms text messages | 2.72 (0.66) |
  Goals text messages | 2.88 (0.33) |
  Protective Behavioral Strategies text messages | 2.48 (0.14) |

4. Secondary Outcome: 6 Week Alcohol Initiation (Number of Participants Who Initiated Drinking)
Description: Number of participants who initiated drinking since the baseline assessment
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 40 | 43
Participants | 6 | 3

5. Secondary Outcome: 3 Month Alcohol Initiation (Number of Participants Who Initiated Drinking)
Description: Number of participants who initiated drinking at the 3 month assessment since the 6 week assessment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 32 | 40
Participants | 4 | 3

6. Secondary Outcome: 6 Month Alcohol Initiation (Number of Participants Who Initiated Alcohol Use)
Description: Number of participants who initiated alcohol use at 6 month assessment since the 3 month assessment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 37 | 44
Participants | 4 | 7

7. Secondary Outcome: 9 Month Alcohol Initiation (Number of Participants Who Initiated Alcohol Use)
Description: Number of participants who initiated drinking at 9 month assessment since the 6 month assessment
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 39 | 44
Participants | 6 | 4

8. Secondary Outcome: 6 Week Alcohol Quantity (Number of Drinks Per Week)
Description: Number of drinks consumed each week as measured at 6 week assessment
Time Frame: 6 weeks
Population: Mean and SD of number of drinks consumed each week using the Daily Drinking Questionnaire
Measure: Mean (Standard Deviation); unit: drinks per week
Groups:
- Text Messaging Intervention Group: Participants in the Text MessagingIntervention condition will be provided a predetermined number of messages per week (based partially on responses from Phase 2 focus group) for 6 weeks delivered on Thursdays, Fridays, and Saturdays, which are the most common days of the week that heavy drinking occurs as well as other days and times that focus group participants indicated would be the most helpful.
  Text Messaging Intervention: The content for the Text Messaging Intervention will be designed to be non-confrontational in tone, seek to increase motivation to drink lightly or not at all, and based both on general information about light and non-drinking as well as information provided during the baseline assessment.
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 40 | 43
drinks per week | 1.89 (2.98) | 2.03 (3.34)

9. Secondary Outcome: 3 Month Alcohol Quantity (Number of Drinks)
Description: Number of drinks consumed each week as measured at 3 month assessment
Time Frame: 3 months
Population: Mean and SD of number of drinks consumed each week using the Daily Drinking Questionnaire
Measure: Mean (Standard Deviation); unit: drinks per week
Groups:
- Active Control: Participants in the assessment only control will not receive any text messages, but will complete all survey assessments on the same schedule as the Text Message Intervention Group.
Arm/Group | Text Messaging Intervention Group | Active Control
Number analyzed (Participants) | 32 | 40
drinks per week | 1.52 (2.38) | 2.03 (2.78)

10. Secondary Outcome: 6 Month Alcohol Quantity (Number of Drinks Consumed Per Week)
Description: Number of drinks consumed each week as measured at 6 month assessment
Time Frame: 6 months
Population: Mean and SD of number of drinks consumed each week using the Daily Drinking Questionnaire
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 37 | 44
drinks per week | 1.48 (2.62) | 1.67 (3.39)

11. Secondary Outcome: 9 Month Alcohol Quantity (Number of Drinks Consumed Per Week)
Description: Number of drinks consumed each week as measured at 9 month assessment
Time Frame: 9 months
Population: Mean and SD of number of drinks consumed each week using the Daily Drinking Questionnaire
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
Number analyzed (Participants) | 39 | 44
drinks per week | 1.46 (2.74) | 1.21 (2.20)

ADVERSE EVENTS:
Time Frame: Data was collected over 9 months.
Description: The definition used is the same as the clinical trials.gov definition.
Arm/Group | Text Messaging Intervention Group | Assessment Only Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

LIMITATIONS AND CAVEATS:
The trial, which studied the Freshman college experience, took place during the COVID-19 pandemic, and thus results may not fully generalize.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03750838/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03750838/SAP_001.pdf